CLINICAL TRIAL: NCT04519034
Title: Retrospective Pilot Study of Vitamin D Status and Immune-inflammatory Status in Different UK Populations With COVID-19 Infection
Brief Title: Vitamin D Status and Immune-inflammatory Status in Different UK Populations With COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 285176
Record Dates: First submitted 2020-08-03; First posted 2020-08-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: vitamin D; cytokines; ethnicity; pro-inflammatory molecules
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Audit 1: All vitamin D results performed since January 2020 (N= ~15000) together with age, weight and height if available, ethnicity and other relevant laboratory markers (Ca, adjusted calcium, PTH, Mg, phosphate, liver and renal profile, Covid-19 screening, CRP, Haematinics, FBC)
  Interventions: Other: no intervention
- Audit 2: All Covid-19 screening results together with vitamin D, ethnicity, age, weight, height, length of stay in hospital including ICU (if applicable), type of illness, recovered or not, associated health conditions, CRP, Ferritin, Haematinics, vitamin A and E, procalcitonin, LDH, INR, fibrinogen, FBC, D-dimers, CK, Troponin-T, cytokines, renal function and electrolytes from patients tested at GSTT NHS Trust.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — There will be no intervention

SUMMARY:
Hypothesis: Serum Vitamin D (25(OH)D) is significantly lower in severe versus non-severe COVID-19 infections and that this is a function of ethnicity. There is an association between vitamin D status and various cytokines (pro-inflammatory molecules).

The primary objective of this research is to provide a snap shot of vitamin D status in patients from the South-East London area by age, sex, ethnicity and BMI and demonstrate ethnic differences in vitamin D status as well as its associations with severe vs non-severe COVID-19 infections.

The secondary objective is to determine if there is an association between vitamin D status and various cytokines (pro-inflammatory molecules) and severity of disease.

DETAILED DESCRIPTION:
Worldwide there has been over 6 million cases and 380,810 deaths from Coronavirus 2019 (COVID-19) (ECDC June 2020). According to the European Centre for Disease Prevention and Control (ECDC) risk factors for critical illness include elderly people above 70 years of age, and people with underlying conditions such as hypertension, diabetes, cardiovascular disease, chronic respiratory disease, immune compromised status and obesity (73.4% of critically ill patients with BMI 30-40). In addition, in the UK 32% of critically ill COVID-19 patients are of Black or Asian ethnic-minority background (ICNARC April 10th, 2020). There is therefore an urgent need to fully understand the risk factors for severe COVID-19 infection and find an effective treatment. In COVID-19 infection those patients that required intensive care treatment have high circulating cytokines and chemokines TNF-α, IL-2, IL-6, IL-7, IL-9, IL-17, IFN-γ, MCP-1 and MIP-1α. Severe COVID-19 infection appears therefore to be associated with a damaging hyperinflammation state. In addition to a dysregulated cytokine response there is also dysregulation of immune cell populations in COVID-19 infection. For example, there is low T regs, NK cell and CD8+ and CD4+ T cells in severe COVID-19 infection. Moreover, CD8+ T cells appear to be an independent predictor for COVID-19 severity and treatment efficacy.

Other than genetic factors, e.g. HLA, which may predispose to severe COVID-19, vitamin D (25(OH)D) may be important for several reasons. Firstly because 25(OH)D inadequacy is prevalent in European and US older adults (>60 years), Black and Asian minority ethnic population groups and in those with a high BMI. Secondly because 25(OH)D is known to have important immunoregulatory roles e.g. in downregulating pro-inflammatory cytokines TNF-α, IL-1, IL-2, IL-6, IL-8, IL-17, IFN-γ and upregulating anti-inflammatory TGFβ and IL-10. 25(OH)D also promotes Treg and effector CD8+ T cell differentiation and expansion. Furthermore, 25(OH)D has a role in preventing and reducing human respiratory infections e.g. influenza and in experimental animals is positively associated with virus specific CD8+ T cells. Vitamin D may also be an important modulator of hyperinflammatory response in patients with Covid-19 infection through cytokine storm suppression.

As part of the Government's response to Covid-19, Public Health England has re-issued existing advice on vitamin D: https://www.nhs.uk/conditions/vitamins-and-minerals/vitamin-d/ This study will provide important information on vitamin D status as a possible risk factor in relation to COVID-19 infection in UK elderly and ethnic minority populations. Furthermore, the data generated could also have important implications for future supplementation and or vaccination strategies for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All patients tested for vitamin D and Covid-19

Exclusion Criteria:

* not applicable

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients tested for vitamin D and Covid-19
Sampling Method: Probability Sample
Enrollment: 27628 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Collecting vitamin D results in patients from the South-East London area together with age, sex, ethnicity and BMI and other relevant laboratory results. | January-June 2020
  All vitamin D results performed by the Nutristasis Unit at St. Thomas' since January 2020 (N= ~15000) together with age, weight and height if available, ethnicity and other relevant laboratory markers (Ca, adjusted calcium, PTH, Mg, phosphate, liver and renal profile, Covid-19 screening, CRP, Haematinics, FBC) if they were tested within two weeks of the sample being measured for vitamin D will be acquired. The results of this audit will provide a snap shot of vitamin D status in patients from the South-East London area by age, sex, ethnicity and BMI (weight in kg/height2). Correlation analysis will also be undertaken with other laboratory parameters.

SECONDARY OUTCOMES:
Collecting Covid-19 screening results together with age, sex, ethnicity and BMI and other relevant laboratory results. | March-June 2020
  All Covid-19 screening results together with vitamin D (nmol/L), ethnicity, age (yrs), weight (m) and height to obtain BMI, length of stay in hospital including ICU in days (if applicable), type of illness, recovered or not (y or no), associated health conditions, CRP, Ferritin, Haematinics, vitamin A and E, procalcitonin, LDH, INR, fibrinogen, FBC, D-dimers, CK, Troponin-T, cytokines, renal function and electrolytes will be collected from patients tested at GSTT NHS Trust.
  We expect that only a small number of patients who had Covid-19 screening performed would have had vitamin D, cytokines and other markers measured. However, we estimate that we will be able to identify a sufficient number of Covid-19 patients for regression and correlation analysis from this data.

CONTACTS AND LOCATIONS:
Overall Officials: Agata Sobczynska-Malefora, PhD, Principal Investigator — GSTT NHS Trust
Locations (1):
- GSTT NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Shen L, Li S, Zhu Y, Zhao J, Tang X, Li H, Xing H, Lu M, Frederick C, Huang C, Wong G, Wang C, Lan J. Clinical and laboratory-derived parameters of 119 hospitalized patients with coronavirus disease 2019 in Xiangyang, Hubei Province, China. J Infect. 2020 Jul;81(1):147-178. doi: 10.1016/j.jinf.2020.03.038. Epub 2020 Apr 10. No abstract available. PMID 32283164
- [Background] Daneshkhah A, Agrawal V, Eshein A, Subramanian H, Roy HK, Backman V. Evidence for possible association of vitamin D status with cytokine storm and unregulated inflammation in COVID-19 patients. Aging Clin Exp Res. 2020 Oct;32(10):2141-2158. doi: 10.1007/s40520-020-01677-y. Epub 2020 Sep 2. PMID 32876941
- [Background] O'Neill LA, Kishton RJ, Rathmell J. A guide to immunometabolism for immunologists. Nat Rev Immunol. 2016 Sep;16(9):553-65. doi: 10.1038/nri.2016.70. Epub 2016 Jul 11. PMID 27396447
- [Background] Surman SL, Jones BG, Woodland DL, Hurwitz JL. Enhanced CD103 Expression and Reduced Frequencies of Virus-Specific CD8+ T Cells Among Airway Lymphocytes After Influenza Vaccination of Mice Deficient in Vitamins A + D. Viral Immunol. 2017 Dec;30(10):737-743. doi: 10.1089/vim.2017.0086. Epub 2017 Nov 13. PMID 29130830
- [Background] Bergman P, Lindh AU, Bjorkhem-Bergman L, Lindh JD. Vitamin D and Respiratory Tract Infections: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. PLoS One. 2013 Jun 19;8(6):e65835. doi: 10.1371/journal.pone.0065835. Print 2013. PMID 23840373
- [Background] Martineau AR, Jolliffe DA, Greenberg L, Aloia JF, Bergman P, Dubnov-Raz G, Esposito S, Ganmaa D, Ginde AA, Goodall EC, Grant CC, Janssens W, Jensen ME, Kerley CP, Laaksi I, Manaseki-Holland S, Mauger D, Murdoch DR, Neale R, Rees JR, Simpson S, Stelmach I, Trilok Kumar G, Urashima M, Camargo CA, Griffiths CJ, Hooper RL. Vitamin D supplementation to prevent acute respiratory infections: individual participant data meta-analysis. Health Technol Assess. 2019 Jan;23(2):1-44. doi: 10.3310/hta23020. PMID 30675873
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- See also: Abstract presented at XII Immunonutrition Conference in — https://www.researchgate.net/publication/353247283_Vitamin_D_deficiency_is_more_common_in_UK_black_people_and_a_possible_COVID-19_risk_factor_Abstract_45151_XII_ISIN_Conference_on_Immunonutrition_July_14-16th_2021_Ann_Nutr_Metab_July_13_2021